CLINICAL TRIAL: NCT03971942
Title: Department of Psychology, Hunan Normal University
Brief Title: Neutral and Positive Attention Bias Modification Training for Young Adults With Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, Wenhui Yang, Department of Psychology, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABM2017
Record Dates: First submitted 2019-03-26; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Depressive Disorder
Keywords: attention bias modification; positive attention bias; depressive symptoms; prevention
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neutral ABMT (Experimental): 8-session-ABMT during a two-week period and 4-session-booster-ABMT during a two-week period
  Interventions: Behavioral: Neutral ABMT
- Positive ABMT (Experimental): 8-session-ABMT during a two-week period and 4-session-booster-ABMT during a two-week period
  Interventions: Behavioral: Positive ABMT

INTERVENTIONS:
Behavioral: Neutral ABMT — In the neutral attention bias, there are 108 pairs of neutral-negative words, 54 pairs of which are used in the training group and 54 pairs of which are used in the placebo group. The word pairs in each group are repeated 4 times, with a total of 216 trial. Participants received 8 sessions over 2 weeks (1 session every other day).In booster ABMT, participants received 4 sessions over 2 weeks (1 session every three days).90% of the targets in the training group appear in the neutral word position and 10% of the targets appear in the negative word position, while 50% of the targets in the placebo group appear in the neutral word position and 50% of the targets appear in the negative word position.
  Arms: Neutral ABMT
Behavioral: Positive ABMT — In the positive attention bias, there are 54 pairs of neutral-negative words, 27 pairs of which are used in the training group and 27 pairs of which are used in the placebo group. The word pairs in each group are repeated 8 times, with a total of 216 trial.Participants received 8 sessions over 2 weeks (1 session every other day). In booster ABMT, participants received 4 sessions over 2 weeks (1 session every three days).90% of the targets in the training group appear in the positive word position and 10% of the targets appear in the neutral word position, while 90% of the targets in the placebo group appear in the neutral word position and 10% of the targets appear in the positive word position.
  Arms: Positive ABMT

SUMMARY:
This study intends to explore the therapeutic effects of the development of negative attention bias modifaction and positive attention bias on depressive symptoms and redundancy through two different attention training methods: (1) neutral attention training (when neutral and sad stimuli are presented simultaneously, attention is always directed towards neutral stimuli to correct negative attention bias) and (2) positive attention training (when neutral and positive stimuli are presented simultaneously, attention is always directed towards positive stimuli to develop positive attention bias).

DETAILED DESCRIPTION:
Attention Bias Modification Training was a modified dot-probe task. In the neutral attention bias, 90% of the targets in the training group appear in the neutral word position and 10% of the targets appear in the negative word position, while 50% of the targets in the placebo group appear in the neutral word position and 50% of the targets appear in the negative word position. In the positive attention bias, 90% of the targets in the training group appear in the positive word position and 10% of the targets appear in the neutral word position, while 90% of the targets in the placebo group appear in the neutral word position and 10% of the targets appear in the positive word position. The investigators assess attention bias scores, depressive symptoms, trait anxiety, rumination and self-report attention control ability at 1-week, 2-week, 4-week, 7-week, 3-month, 4-month, 5-month, 6-month and 12-month follow-ups after training.

ELIGIBILITY:
Inclusion Criteria:

* A score of 14 or higher on the Beck Depression Inventory-Ⅱ

Exclusion Criteria:

1. a current episode of MDD, bipolar disorder, schizophrenia or organic mental disorder;
2. any concurrent psychotherapy;
3. any concurrent psychotropic medication.

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2017-12-24 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Changes of attentional bias score | pre-training, post-training(2 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month( booster pre-training), 4-month (booster post-training), 5-month,6-month,12-month after post-training)
  Attentional bias score tested by a typical dot-probe task
Changes of depressive symptoms | pre-training, post-training(2 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month( booster pre-training), 4-month (booster post-training), 5-month,6-month,12-month after post-training)
  Depression symptoms tested by clinicians using the Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children (K-SADS)

SECONDARY OUTCOMES:
Changes of self-reported depressive symptoms | pre-training, post-training(2 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month( booster pre-training), 4-month (booster post-training), 5-month,6-month,12-month after post-training)
  Self-reported depressive symptoms assessed by Beck depression scale-second version (BDI-II)
Changes of self-reported rumination | pre-training, post-training(2 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month( booster pre-training), 4-month (booster post-training), 5-month,6-month,12-month after post-training)
  Self-reported rumination assessed by Rumination Response Scale(RRS).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Hunan Normal University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code